CLINICAL TRIAL: NCT05676164
Title: A Multicenter, Prospective, Randomized Controlled Clinical Study to Evaluate the Safety and Efficacy of Oral Contrast Agent for Sonography
Brief Title: A Study to Evaluate the Safety and Efficacy of Oral Contrast Agent for Sonography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong Branden Med.Device Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: B202103
Record Dates: First submitted 2022-12-01; First posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-12

CONDITIONS: Unspecified Disorder of Stomach and Duodenum

STUDY DESIGN:
Intervention Model Description: A Multicenter, Prospective, Randomized Controlled Clinical Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Oral Contrast Agent for Sonography from Huzhou East Asia Medical Supplies Co., LTD
  Interventions: Device: TIAN XIA
- Experimental group (Experimental): Oral Contrast Agent for Sonography from Shandong branden Medical Device Co., LTD
  Interventions: Device: KANG XIAN

INTERVENTIONS:
Device: KANG XIAN — This product is a liquid composed of silica, stabilizer, xylitol, flavoring agent and water. The pH value of the product is 5.0 ~ 8.0, and the total heavy metal content (measured by Pb2+) is less than 10µg/ml.
  Arms: Experimental group
Device: TIAN XIA — The products are dark yellow granules made from rice, soybean, lotus root powder, orange peel, coix seed and yam.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to verify the safety and efficacy of Oral Contrast Agent for Sonography produced by Shandong Baiduo Medical Instruments Co., LTD.

DETAILED DESCRIPTION:
The goal of this clinical trial is to verify the safety and efficacy of Oral Contrast Agent for Sonography produced by Shandong Baiduo Medical Instruments Co., LTD.

Participants will Ultrasound was administered with Oral Contrast Agent for Sonography and observed for 2 days.

The investigators will compare Oral Contrast Agent for Sonography produced by Huzhou East Asia Medical Supplies Co., LTD to see if the safety and efficacy of Oral Contrast Agent for Sonography produced by Shandong Baiduo Medical Instruments Co., LTD

ELIGIBILITY:
Inclusion Criteria:

1. subjects whose physicians recommend oral gastrointestinal CEUS;
2. subjects aged 18-80 years;
3. The subject or guardian can understand the purpose of the study, voluntarily sign the informed consent, and agree to the clinical follow-up;

Exclusion Criteria:

1. Pregnant and lactating women;
2. Subjects with dysphagia;
3. Subjects suspected of gastric bleeding, gastrointestinal perforation, intestinal disorders or gastrointestinal obstruction;
4. Subjects who are expected to receive surgery within 60 hours;
5. Subjects who have received gastroscopy within 24 hours;
6. subjects deemed unsuitable for the study by the researcher;
7. Subjects who have participated in other drug or device clinical trials and have not completed the expected primary endpoint follow-up of the clinical trials in which they participated.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
Ultrasonic display rate of stomach and duodenal bulb | 1 hour ± 0.5 hour after examination
  The grade evaluation of the display effect will be determined by the total score of the gastric wall hierarchy and structure, the stomach and duodenal bulb morphology evaluation: 0-2 points for poor, 3-4 points for average, and 5-6 points for excellent. The total score of the display effect is greater than 2 points. After the end of the experiment, the sum of the number of cases with average and excellent imaging is divided by the total number of cases, and then multiplied by 100%, which is the ultrasonic display rate of the stomach and duodenal bulb.

SECONDARY OUTCOMES:
Anti-interference capability of product | 1 hour ± 0.5 hour after examination
  The satisfaction degree of the product's anti-interference ability refers to the satisfaction degree of the doctor's observation of the product in the stomach and duodenal bulb of the subject due to the product's homogeneity and the ability to eliminate gas artifacts.
Stomach filling and peristaltic emptying | 1 hour ± 0.5 hour after examination
  Stomach filling and peristaltic emptying represent the condition of stomach filling and peristaltic emptying observed by the study physician.
Ease of operation | 1 hour ± 0.5 hour after examination
  Ease of operation refers to the time required to prepare the device before use by the subject. The shorter the time, the better the ease of operation.
Incidence of device adverse events | 48 hours ±12 hours after examination
  Device adverse events refer to device-related nausea, vomiting, abdominal pain, diarrhea, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Huixiong Xu, Dr., Study Chair — Shanghai 10th People's Hospital
Locations (1):
- Qilu Hospital Of Shangdong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No